CLINICAL TRIAL: NCT02443649
Title: Improving Sleep Quality in People With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Barry S. Oken, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB#10810
Record Dates: First submitted 2015-03-10; First posted 2015-05-14 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Primary Insomnia; Psychophysiological Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep hypnosis plus sleep hygiene (Experimental): Those randomized into this group will receive the sleep hygiene program plus hypnosis.
  Interventions: Behavioral: Sleep hygiene program; Behavioral: Sleep hypnosis
- Sleep hygiene only (Active Comparator): Those randomized into this group will receive the Optimizing Sleep Hygiene program during the intervention visit and hypnosis recording after the follow-up visit.
  Interventions: Behavioral: Sleep hygiene program

INTERVENTIONS:
Behavioral: Sleep hygiene program — Sleep hygiene program
Behavioral: Sleep hypnosis — Hypnosis recording with personalized goals and imagery for sleep improvement
  Other Names: Hypnosis
  Arms: Sleep hypnosis plus sleep hygiene

SUMMARY:
Insomnia is a significant problem affecting 10 to 20% of US population. Long-term pharmacological treatments are not recommended due to side effects, with therapy and sleep hygiene education often employed as alternatives. Use of mind-body approaches for insomnia is increasing. One of the most promising mind-body approaches for alleviating sleep problems is hypnosis. Research indicates significant beneficial effects of hypnosis on sleep, but sleep was rarely assessed as primary outcome and studied populations were diverse. Further, it remains unclear who the best candidates for benefitting from hypnosis are. To address some of the gaps in the current knowledge, the study evaluates whether 1) an addition of hypnotic suggestion for sleep improvement to the optimizing sleep hygiene (OSH) program increases the effectiveness of the OSH using objective and subjective assessments and 2) determines characteristics associated with hypnotic responsiveness.To address these goals a randomized controlled trial (RCT) with 3 laboratory visits (baseline, intervention, and 1 month follow-up) will be conducted with 50 adults meeting criteria for primary insomnia and allocated to one the two groups: 1) experimental group receiving during the intervention visit a combination of the Optimizing Sleep Hygiene (OSH) program and a hypnosis session for sleep improvement and 2) a control group receiving at the intervention visit the OSH only. Hypnosis session for sleep improvement for the control group will be offered at the end of the follow-up study visit (conducted after 4 weeks post-intervention) after completing all follow-up measures. Each study visit will last for 2-3 hours. During the visits sleep, personality traits and daily function of the participants will be assessed. Further, after the baseline and one week before the follow-up visit subjects will wear a watch-like actigraphic device monitoring their sleep patterns at home and will complete sleep diary.

The knowledge gained from this study will inform the literature and clinicians about usefulness of hypnosis for insomnia sufferers and will help identify the population of insomnia sufferers most likely benefit from use of hypnosis for sleep

DETAILED DESCRIPTION:
1. Protocol Title Improving sleep quality in people with insomnia
2. Objectives The purpose of the study is to compare effectiveness of two sleep improvement programs for people with primary psychophysiological insomnia: 1) the Optimizing Sleep Hygiene (OSH) program and 2) a combination of the OSH and hypnosis for sleep improvement. The goals of this study are: 1) using objective and subjective assessments to evaluate whether an addition of hypnotic suggestion for sleep improvement to the sleep hygiene program increases the effectiveness of the OSH, and 2) to determine subject characteristics associated with hypnotic responsiveness in adults with primary psychophysiological insomnia.

   To address these goals a randomized controlled trial (RCT) with 3 laboratory visits (baseline, intervention, and 1-month follow-up) will be conducted with 50 adults meeting criteria for psychophysiological insomnia and allocated to one the two groups: 1) experimental group receiving during the intervention visit a combination of the Optimizing Sleep Hygiene (OSH) program and a hypnosis session for sleep improvement and 2) a control group receiving at the intervention visit the OSH only. One-month follow-up visit will be conducted following at least 4 weeks since the intervention visit. Hypnosis session for sleep improvement for the control group will be offered at the end of the follow-up study visit after completing all follow-up measures. Each study visit will last for 2-3 hours. During the visits participants' personality traits, hypnotic susceptibility as well as measures of insomnia severity, sleep quality, hygiene, and daily function will be assessed. Further, between the visits at home subjects will wear a watch-like actigraphic device monitoring their day and night activity. These actigraphic recordings will allow for collecting objective actigraphic measures of sleep. The actigraphic measures will be collected along with daily sleep and medications diaries for periods of 7 days immediately after the baseline assessment and 1 week prior to one-month follow-up assessment. Additionally, during the one-month follow-up visit, patterns of brain activity will be monitored in all subjects first when they listen to a neutral sleep-related recording and then during listening to a recording of hypnosis for sleep improvement. The purpose of these measures is to compare brain activity patterns and identify specific biomarkers of hypnotic state. Four weeks after the completion of all study visits participants will provide information about their sleep and their experiences with the study interventions components via a telephone or on-line assessment depending on their choice.The knowledge gained from this study will inform the literature and clinicians about usefulness of hypnosis for insomnia sufferers and will help identify the population most likely benefit from use of hypnosis for sleep. The goals of the proposal will be addressed by the following specific aims:

   Specific Aim 1: Compare changes from baseline in sleep parameters at the one-month follow-up visit between the two study groups (experimental and control) after exposure to the interventions.

   Hypothesis: Greater improvements in actigraphic and subjective sleep parameters and daily function will be observed in the experimental group compared to the control group.

   Specific Aim 2a: Identify characteristics correlating with changes in measures of sleep quality to describe a population that can potentially benefit from hypnosis.

   Hypothesis: Several sleep-specific variables (e.g. specific baseline insomnia symptoms and sleep hygiene problems) and personality features (e.g. hypnotic susceptibility and specific personality traits) will correlate with post-intervention changes in sleep variables.

   Specific Aim 2b: Identify characteristics correlating with hypnotic susceptibility for creating a scale that can be used in a clinic to assess hypnotic responsiveness for sleep-related problems.

   Hypothesis: Using the items from the instruments given during the study identified as a part of Specific Aim 2a short instrument could be constructed that can quickly and reliably categorize people based on their hypnotic responsiveness for sleep-related problems.

   Specific Aim 3: Assess brain wave patterns concurrent with hypnosis to identify psychophysiological markers specific to hypnotic state in order to describe mechanisms underlying hypnosis.

   Hypothesis: Based on the differences between the two states: 1) listening to hypnosis and 2) listening to a neutral sleep-related recording, brain activity markers that can distinguish state of hypnosis from the state of listening to a neutral recording could be identified.

   Background Insomnia, characterized by non-restorative sleep or by difficulty in initiating or maintaining sleep, is a significant problem affecting 10 to 20% of US population. Poor sleep impairs cognitive and immune functions, mood and productivity of sufferers and can increase risk for hypertension, diabetes, cancer and overall mortality. Long-term pharmacological insomnia treatment is not recommended due to side effects, with therapy and sleep hygiene education often employed as alternatives. There is also a growing interest in using mind-body approaches for managing sleep problems. Mind-body approaches are becoming popular due to accessibility and low side effect profile, as well as due to increasing amount of research evidence indicating their effectiveness. For example, a recent review of mind-body methods for improving sleep revealed that among the most promising mind-body approaches for alleviating sleep problems was hypnosis. Hypnosis is a state of relaxation combined with highly focused attention and characterized by dissociation of competing thoughts and sensations towards the periphery of awareness. One way to achieve hypnotic state is through an induction procedure typically followed by hypnotic suggestions or statements intended to elicit behavioral change. Efficacy of hypnosis has been demonstrated for several conditions, most notably for decreasing pain and alleviating stress-related disorders. Using hypnosis for sleep improvement is still a developing area of research. Though several studies found significant beneficial effects of hypnosis on sleep, most studies used hypnosis for alleviating other problems influencing sleep (e.g. hot flashes) rather than specifically targeting sleep as the primary focus of improvement. Moreover, majority of the studies on sleep and hypnosis used only subjective measures for evaluating sleep quality. Further, it remains unclear who the best candidates for benefitting from hypnosis are and how hypnotic responsiveness can be assessed in a clinic without lengthy tests of hypnotic susceptibility. To address some of the gaps in the current knowledge, the goals of this study are: 1) using objective and subjective assessments to evaluate whether an addition of hypnotic suggestion for sleep improvement to the sleep hygiene education program increases the program effectiveness, and 2) to determine subject characteristics associated with hypnotic responsiveness in adults with primary psychophysiological insomnia.
3. Design: The planned study is a single-blind two-arm randomized controlled trial (RCT) with three study visits (baseline, intervention, and one-month follow-up), with participants randomly assigned to receive Optimizing Sleep Hygiene (OSH) program as an intervention either alone or in conjunction with hypnosis for sleep improvement during the intervention visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 or older
* Primary insomnia diagnosis
* Able to attend all study sessions and willing to complete the study requirements
* Fluent English
* Able and willing to consent

Exclusion Criteria:

* Current use of hypnosis with hypnotist
* Other diagnosed sleep disorders
* Other serious illness (e.g. cancer, major depression, chronic pain condition etc.)
* Problem hearing
* Pregnancy
* Use of illicit drugs or alcohol use in excess of what constitutes moderate drinking (>1 drink per day for women and >2 drinks per day for men)

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency change at one-month follow-up (from baseline) | collected at baseline and one-month follow-up
  actigraphic sleep efficiency

SECONDARY OUTCOMES:
Functional outcomes of sleep score change at one-month follow-up (from baseline) | collected at baseline and one-month follow-up
  Functional outcomes of sleep score collected at baseline and follow-up through FOSQ
Sleep Hygiene score change at one-month follow-up (from baseline) | collected at baseline and one-month follow-up
  Sleep Hygiene Index instrument score

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Oken, MD, MS, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States